CLINICAL TRIAL: NCT01267292
Title: Psychopharmacology of Novel Medications for Cocaine Dependence - Buspirone
Brief Title: Psychopharmacology for Cocaine Dependence - Buspirone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Scott Lane, Professor - Psychiatry & Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NIDA-P50-09262-Project2.1
Record Dates: First submitted 2010-12-24; First posted 2010-12-28 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; psychopharmacology; attentional bias; risky decision making; buspirone; methylphenidate
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Buspirone; Starch; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buspirone plus Methylphenidate (Experimental): [week 1: Buspirone 30 mg twice a day (9am and 6pm) on Monday through Sunday; no Methylphenidate or Methylphenidate placebo] [week 2: Buspirone 45 mg twice a day (9am and 6pm) on Monday through Sunday; 0mg Methylphenidate (placebo) on Monday at 10am; Methylphenidate once a day (10am) on Wednesday and Friday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)] [week 3: Buspirone 45 mg twice a day (9am and 6pm) on Monday through Sunday; Methylphenidate once a day (10am) on Monday and Wednesday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)]
  Interventions: Drug: Buspirone; Drug: Methylphenidate; Drug: Placebo for Methylphenidate
- Placebo for Buspirone plus Methylphenidate (Placebo Comparator): [week 1: Placebo for Buspirone twice a day (9am and 6pm) on Monday through Sunday; no Methylphenidate or Methylphenidate placebo] [week 2: Placebo for Buspirone twice a day (9am and 6pm) on Monday through Sunday; 0mg Methylphenidate (placebo for Methylphenidate) on Monday at 10am; Methylphenidate once a day (10am) on Wednesday and Friday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)] [week 3: Placebo for Buspirone twice a day (9am and 6pm) on Monday through Sunday; Methylphenidate once a day (10am) on Monday and Wednesday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)]
  Interventions: Drug: Placebo for Buspirone; Drug: Methylphenidate; Drug: Placebo for Methylphenidate

INTERVENTIONS:
Drug: Buspirone — [week 1: Buspirone 30 mg twice a day (9am and 6pm) on Monday through Sunday] [weeks 2-3: Buspirone 45 mg twice a day (9am and 6pm) on Monday through Sunday]
  Other Names: Buspar
  Arms: Buspirone plus Methylphenidate
Drug: Placebo for Buspirone — [week 1: Placebo for Buspirone twice a day (9am and 6pm) on Monday through Sunday] [weeks 2-3: Placebo for Buspirone twice a day (9am and 6pm) on Monday through Sunday]
  Other Names: corn starch
  Arms: Placebo for Buspirone plus Methylphenidate
Drug: Methylphenidate — Methylphenidate serves as an acute stimulant challenge. [week 1: no Methylphenidate or Methylphenidate placebo] [week 2: 0mg Methylphenidate (placebo for Methylphenidate) on Monday at 10am; Methylphenidate once a day (10am) on Wednesday and Friday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)] [week 3: Methylphenidate once a day (10am) on Monday and Wednesday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)]
  Other Names: Ritalin
Drug: Placebo for Methylphenidate — [week 1: no Methylphenidate or Methylphenidate placebo] [week 2: 0mg Methylphenidate (placebo for Methylphenidate) on Monday at 10am; Methylphenidate once a day (10am) on Wednesday and Friday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)] [week 3: Methylphenidate once a day (10am) on Monday and Wednesday, and on each of these 2 days the Methylphenidate dose will be different (15 mg, 30mg, 60 mg, or 0mg)]
  Other Names: corn starch

SUMMARY:
Chronic cocaine use may produce disruption of neurotransmitter functions (including dopamine). This may in turn contribute to measurable dysfunction in important cognitive and behavioral processes. Stimulants that enhance dopamine (DA) function may help in treating cocaine dependence and improving behavioral function -- supporting the notion that these processes are related. An important step is to understand the subjective, physiological, and behavioral effects of potential medications for cocaine dependence.

DA-modulating drugs may be targets for pharmacotherapy for substance dependence, and particularly for stimulant drugs like cocaine, which disrupt normal DA function. Buspirone is currently the only available dopamine subtype 3 (DA3) approved for human administration, and is thus a viable investigational compound.

This project proposes to evaluate the DA-modulating effects of buspirone on behavioral deficiencies related to DA depletion. Accordingly, the project aims to characterize the effects of buspirone in individuals with cocaine dependence. Employing a daily dosing designs within an acute stimulant challenge (methylphenidate), the experiment will characterize the subjective effects, cardiovascular effects, and behavioral effects (attentional bias to drug cues and risky decision making). The primary hypotheses are that buspirone will attenuate the increases in subjective drug effects ("stimulated", "like drug") and behavioral effects (increases in attentional bias and risky decision making) that are produced by acute methylphenidate administration.

DETAILED DESCRIPTION:
Chronic cocaine use may produce disruption of monoamine systems (including dopamine). This may in turn contribute to measurable dysfunction in important cognitive and behavioral processes. Pharmacotherapy with stimulants that enhance dopamine (DA) function has shown efficacy in treating cocaine dependence and improving behavioral function -- supporting the notion that these processes are related. In the development of novel pharmacotherapies for cocaine dependence, an important step is a full characterization of the psychopharmacological properties of potential medications for cocaine dependence, including subjective, physiological, and behavioral effects. Selective medications may play a key role in the modulation of DA neurotransmission by enhancing DA receptor activation.

The D3 receptor is an autoreceptor that may function to control phasic DA activity and mediate sensitization of DA agonists, thus playing a role in conditioning of drugs of abuse like cocaine. Growing evidence suggests that D3 receptor antagonists may be targets for pharmacotherapy for substance dependence, and particularly for stimulant drugs like cocaine, which disrupt normal DA function. Importantly, administration of D3 antagonists may disrupt reactivity (attention) to drug cues and attenuate cue-induced craving. Buspirone is currently the only available D3 antagonist approved for human administration, and is thus a viable investigational compound.

This project proposes to evaluate the potential pharmacotherapeutic action of the D3 antagonist buspirone. The DA-modulating effects of buspirone may help with affective and behavioral deficiencies related to DA depletion. Accordingly, the project aims to characterize the psychopharmacology of buspirone in individuals with cocaine dependence. Employing chronic dosing designs within an acute stimulant challenge (methylphenidate), the experiment will be conducted using well-established psychopharmacological methods in order to characterize the shape and magnitude of chronic pretreatment-mediated change in the methylphenidate dose-response curve. Measures will include subjective effects, cardiovascular effects, and behavioral effects (attentional bias to drug cues and risky decision making). These data will compliment and provide valuable information to clinical trials using these agents to treat cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* cocaine dependent subjects, non-treatment seeking
* meet current DSM-IV criteria for cocaine dependence disorder
* report using cocaine within the past 30 days
* at least 1 positive urine toxicology screen for the cocaine metabolite benzoylecgonine (BE) [300 ng/mL, during the initial (2-4 day) screening period
* acceptable health on the basis of interview, medical history, and physical exam
* able to understand the consent form and provide written informed consent.

Exclusion Criteria:

* currently dependent on any psychoactive substance other than cocaine or nicotine
* current DSM-IV diagnosed major psychiatric disorder (e.g., psychosis, bipolar, major depressive disorder)
* any medical condition that would contraindicate administration of medications
* taking medications known to have significant drug interactions study medications
* probation / parole requiring reports of drug use to court officers
* pregnant or nursing for female patients
* cannot read, write, or speak English.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lane, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Started | 24 | 26
Completed | 20 | 20
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (7.82) | 44.15 (7.23) | 42.925 (7.525)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Attentional Bias as assessed by score on the Stroop task [Mean (Standard Deviation); unit: milliseconds] — The baseline reading was assessed on Monday of week 2. Participants are instructed to respond to words shown in different colors on the screen by pressing as quickly and accurately as possible on one of three colored buttons. Attentional bias is measured as the difference in reaction times on cocaine vs. neutral words. The reported score is a difference score in milliseconds (cocaine minus neutral), in which positive means slower to respond to cocaine and thus greater attentional bias, and negative means no attentional bias to cocaine words.
  milliseconds | 12.39759 (70.25051) | 28.67933 (69.99501) | 20.53846 (70.12276)
Risky decision making as assessed by score on the risky decision making task [Mean (Standard Deviation); unit: units on a scale] — The baseline reading was assessed on Monday of week 2. The risky decision making task provides subjects with three choice options on each of 100 repeated trials. Options are low, moderate, and high risk, based on variance and probability in gain/loss amounts. The low risk option is more adaptive over many trials. The outcome measure is a risk index (ranging from 0.33 to 100) that factors in tolerance for variability and amount of gains and losses across the three options. 100 is highest risk. 0.33 is lowest risk.
  units on a scale | 9.778235 (7.368139) | 8.945935 (5.512101) | 9.362085 (6.44012)
Subjective Effects as assessed by score on the Vigor Subscale of the Profile of Mood States (POMS) [Mean (Standard Deviation); unit: units on a scale] — The baseline reading was assessed on Monday of week 2. The POMS is a self-rating measure of current mood, consisting of six subscales demonstrated to be sensitive to a range of acute drug effects, including amphetamine, cocaine, and caffeine. A 37-item short form of the POMS was used, which correlates highly with the full scale. The vigor subscale is reported, and the vigor subscale score ranges from 0 to 28, with 28 representing the highest score for that mood state. The higher the value, the worse the outcome.
  units on a scale | 5.989247 (6.306573) | 5.080925 (5.594259) | 5.535086 (5.950416)
Subjective Effects as assessed by Score on "Feel High" Subscale of the Drug Effects Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The baseline reading was assessed on Monday of week 2. The DEQ is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", "Like Drug", and "Want More". The "Feel High" subscale is reported, and this subscale is scored on a visual analogue scale (scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
  units on a scale | 15.32065 (25.31205) | 8.128655 (17.20622) | 11.7246525 (21.259135)
Subjective Effects as assessed by the "elated" subscale of the visual analogue scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The baseline reading was assessed on Monday of week 2. The VAS presents 100-mm horizontal lines labeled with an adjective: "stimulated", "high", "anxious", "elated", "hungry", and "nauseated." The "elated" subscale is reported, and this sub scale is anchored by "not at all" (0) on the left and "extremely" (100) on the right, with a score range of 0-100. The higher the score, the worse the outcome.
  units on a scale | 22.00538 (26.22491) | 20.4593 (26.25991) | 21.23234 (26.24241)
Heart rate [Mean (Standard Deviation); unit: beats per minute] — The baseline reading was assessed on Monday of week 2. Heart rate is the measure of heart beats per minute.
  beats per minute | 65.42781 (11.223) | 64.44886 (11.28527) | 64.938335 (11.254135)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — The baseline reading was assessed on Monday of week 2. Systolic blood pressure is the amount of pressure in the arteries during contraction of the heart muscle.
  mmHg | 117.4813 (14.13086) | 113.2727 (11.94963) | 115.377 (13.040245)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — The baseline reading was assessed on Monday of week 2. Diastolic blood pressure is the blood pressure when the heart muscle is between beats.
  mmHg | 74.52406 (8.30489) | 75.34091 (8.234265) | 74.932485 (8.2695775)

OUTCOME MEASURES:

1. Primary Outcome: Attentional Bias as Assessed by Score on the Stroop Task
Description: The mean score over all 4 time points is reported in this outcome measure (i.e., a summary score is reported). Each subject contributed 1 data point for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 20 data points per dose level per arm.
  The Stroop task assesses attentional biases to cocaine-related (drug-related) and rewarding (non-drug related) stimuli vs. neutral stimuli. Participants are instructed to respond to words shown in different colors on the screen, by pressing as quickly and accurately as possible on one of three colored buttons. Attentional bias is measured as the difference in reaction times on cocaine vs. neutral words. The reported score is a difference score in milliseconds (cocaine minus neutral), in which positive means slower to respond to cocaine and thus greater attentional bias, and negative means no attentional bias to cocaine words.
Time Frame: 1 time a day on Wednesday and Friday of week 2; 1 time a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
milliseconds
  15 mg methylphenidate | -13.90333 (62.76434) | 27.118 (58.84988)
  30 mg methylphenidate | -9.361269 (30.66139) | 15.35407 (66.51272)
  60 mg methylphenidate | 15.59167 (142.0095) | 23.28063 (42.25839)
  0 mg methylphenidate | 4.688844 (30.59728) | 41.22625 (74.82985)

2. Primary Outcome: Risky Decision Making as Assessed by Score on the Risky Decision Making Task
Description: The mean score over all 4 time points is reported in this outcome measure (i.e., a summary score is reported). Each subject contributed 1 data point for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 20 data points per dose level per arm.
  The risky decision making task provides subjects with three choice options on each of 100 repeated trials. Options are low, moderate, and high risk, based on variance and probability in gain/loss amounts. The low risk option is more adaptive over many trials. The outcome measure is a risk index (ranging from 0.33 to 100) that factors in tolerance for variability and amount of gains and losses across the three options. 100 is highest risk. 0.33 is lowest risk.
Time Frame: 1 time a day on Wednesday and Friday of week 2; 1 time a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
units on a scale
  15mg Methylphenidate | 9.126667 (5.094545) | 10.07396 (5.44448)
  30mg Methylphenidate | 10.77167 (6.58645) | 9.699333 (6.334753)
  60mg Methylphenidate | 8.946263 (6.947867) | 7.889825 (5.277534)
  0mg Methylphenidate | 11.415 (6.147164) | 8.715333 (6.34345)

3. Secondary Outcome: Subjective Effects as Assessed by the Addiction Research Center Inventory (ARCI)
Description: The ARCI short form will be used. It is a 49-item true / false questionnaire that has been empirically-derived to assess five different factors, including euphoria, sedation, and dysphoria. The PCAG scale has proven to be a sensitive measure of subjective effects in many studies administering stimulant drugs.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Population: ARCI data were not collected.
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Subjective Effects as Assessed by Score on the Vigor Subscale of the Profile of Mood States (POMS)
Description: The mean score over all 44 time points is reported in this outcome measure (i.e., the summary score is reported). Each subject contributed 11 data points for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 220 data points per dose level per arm.
  The POMS is a self-rating measure of current mood, consisting of six subscales demonstrated to be sensitive to a range of acute drug effects, including amphetamine, cocaine, and caffeine. The six subscales are: depression, vigor, confusion, tension, anxiety, and fatigue. A 37-item short form of the POMS was used, which correlates highly with the full scale. The vigor subscale is reported, and the vigor subscale score ranges from 0 to 28, with 28 representing the highest score for that mood state. The higher the value, the worse the outcome.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
units on a scale
  15mg Methylphenidate | 4.609626 (5.775599) | 3.770115 (4.558423)
  30mg Methylphenidate | 9.924324 (6.630357) | 6.268571 (5.721696)
  60mg Methylphenidate | 4.745946 (5.702335) | 5.874286 (5.866932)
  0mg Methylphenidate | 6.16129 (6.520306) | 5.735632 (5.360873)

5. Secondary Outcome: Subjective Effects as Assessed by Score on the "Feel High" Subscale of the Drug Effects Questionnaire (DEQ)
Description: The mean score over all 44 time points is reported in this outcome measure (i.e., the summary score is reported). Each subject contributed 11 data points for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 220 data points per dose level per arm.
  The DEQ is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug," "Feel High," "Like Drug," and "Want More." The "Feel High" subscale is reported, and this subscale is scored on a visual analogue scale (scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
units on a scale
  15mg Methylphenidate | 9.322581 (17.49543) | 9.178161 (17.58439)
  30mg Methylphenidate | 12.71351 (22.32222) | 10.78857 (17.63701)
  60mg Methylphenidate | 5.886486 (15.6564) | 9.846591 (20.80863)
  0mg Methylphenidate | 10.39785 (17.27747) | 4.508671 (13.15631)

6. Secondary Outcome: Subjective Effects as Assessed by the "Elated" Subscale of the Visual Analogue Scale (VAS)
Description: The mean score over all 44 time points is reported in this outcome measure (i.e., the summary score is reported). Each subject contributed 11 data points for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 220 data points per dose level per arm.
  The VAS presents 100-mm horizontal lines labeled with an adjective: "stimulated," "high," "anxious," "elated," "hungry," and "nauseated." The "elated" subscale is reported, and this sub scale is anchored by "not at all" (0) on the left and "extremely" (100) on the right, with a score range of 0-100. The higher the score, the worse the outcome.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
units on a scale
  15mg Methylphenidate | 11.48128 (21.53051) | 19.53448 (23.74495)
  30mg Methylphenidate | 28.72973 (29.45967) | 21.42045 (25.17651)
  60mg Methylphenidate | 14.54595 (24.1708) | 21.81143 (27.00221)
  0mg Methylphenidate | 21.95676 (25.58082) | 14.89017 (25.46919)

7. Secondary Outcome: Heart Rate
Description: The mean score over all 44 time points is reported in this outcome measure (i.e., the summary score is reported). Each subject contributed 11 data points for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 220 data points per dose level per arm.
  Heart rate is the measure of heart beats per minute.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
beats per minute
  15mg Methylphenidate | 66.84492 (13.48406) | 67.75568 (14.40208)
  30mg Methylphenidate | 66.43316 (13.03261) | 68.26136 (12.89296)
  60mg Methylphenidate | 66.36364 (10.55586) | 69.13068 (13.71256)
  0mg Methylphenidate | 63.21925 (9.372807) | 69.60795 (12.09863)

8. Secondary Outcome: Systolic Blood Pressure
Description: The mean score over all 44 time points is reported in this outcome measure (i.e., the summary score is reported). Each subject contributed 11 data points for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 220 data points per dose level per arm.
  Systolic blood pressure is the amount of pressure in the arteries during contraction of the heart muscle.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
mmHg
  15mg Methylphenidate | 118.0856 (11.56065) | 115.9205 (9.891666)
  30mg Methylphenidate | 114.8396 (10.86901) | 120.4545 (12.3153)
  60mg Methylphenidate | 114.3904 (12.69334) | 113.6932 (10.50046)
  0mg Methylphenidate | 114.7914 (12.56828) | 115.6932 (10.68976)

9. Secondary Outcome: Diastolic Blood Pressure
Description: The mean score over all 44 time points is reported in this outcome measure (i.e., the summary score is reported). Each subject contributed 11 data points for each dose level of Methylphenidate (15mg, 30mg, 60mg, or 0mg), resulting in a total of 220 data points per dose level per arm.
  Diastolic blood pressure is the blood pressure when the heart muscle is between beats.
Time Frame: 11 times a day on Wednesday and Friday of week 2; 11 times a day on Monday and Wednesday of week 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
mmHg
  15mg Methylphenidate | 74.72727 (8.177168) | 76.71591 (6.985616)
  30mg Methylphenidate | 74.56684 (8.160986) | 78.53409 (8.962077)
  60mg Methylphenidate | 73 (9.153999) | 75.5625 (7.56583)
  0mg Methylphenidate | 72.92513 (9.052699) | 76.88636 (7.938955)

10. Secondary Outcome: Rapid Response Inhibition as Assessed by the Immediate Memory Task (IMT)
Description: Subjects are required to respond selectively to a series of stimuli (e.g., numbers) presented briefly for 500 ms with a 500 ms intertrial interval (ITI). Increases in false alarm rates are interpreted as failures in response inhibition. Five digit numbers are presented on a computer screen every 500 ms sec. Subjects are instructed to respond when the first number of a set was repeated. A "hit" response is scored when a subject correctly responds. Distracters consist of five-digit numbers that are completely different from the first, and numbers in which four of the five digits match the original, with the non-matching number occurring randomly across the five digit places. A response to the number with 4 of 5 digits correct is scored as a "false alarm." The a-prime value reflects the ability of the participant to discriminate between signal (Go stimulus) and noise (No-Go stimulus) and ranges from 0.5 (chance level) to 1 (perfect discrimination).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: a-prime
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
a-prime | 0.8327941 (0.1418202) | 0.8498438 (0.0854399)

11. Secondary Outcome: Rapid Response Inhibition as Assessed by the Immediate Memory Task (IMT)
Description: as for outcome 10
Time Frame: Thursday of week 1
Measure: Mean (Standard Deviation); unit: a-prime
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
a-prime | 0.8673529 (0.0764632) | 0.8551562 (0.0849648)

12. Secondary Outcome: Rapid Response Inhibition as Assessed by the Immediate Memory Task (IMT)
Description: as for outcome 10
Time Frame: Monday of week 4
Measure: Mean (Standard Deviation); unit: a-prime
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
a-prime | 0.8569118 (0.0773489) | 0.8695347 (0.0723827)

13. Secondary Outcome: Reversal Learning as Assessed by Number of Perseverative Errors on the Reversal Learning Task
Description: The task is a rapid-presentation, probablistic gain/loss design. Reversal learning is assessed by means of a simple computerized card game. The paradigm utilizes a visual discrimination task where subjects have to learn to respond to outcome contingencies between two stimuli (high probability gain/low probability loss vs. low probability gain/high probability loss). At an unsignaled time point halfway into testing, the contingencies are reversed; the losing card becomes the winning card and the winning card becomes the losing one. Visual feedback regarding win or loss ($0.20) is provided after each trial and the cumulative total gained/lost is also shown. Using trial-and-error feedback, subjects have to discover which of the two patterns is correct and are instructed to win as much money as possible. The duration of the task is approximately 10 minutes, consisting of 80 trials.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: number of perseverative errors
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
number of perseverative errors | 14.41176 (8.155204) | 10.625 (8.023923)

14. Secondary Outcome: Reversal Learning as Assessed by Number of Perseverative Errors on the Reversal Learning Task
Description: as for outcome 13
Time Frame: Thursday of week 1
Measure: Mean (Standard Deviation); unit: number of perseverative errors
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
number of perseverative errors | 11.78154 (12.04489) | 14.13049 (15.27429)

15. Secondary Outcome: Reversal Learning as Assessed by Number of Perseverative Errors on the Reversal Learning Task
Description: as for outcome 13
Time Frame: Monday of week 4
Measure: Mean (Standard Deviation); unit: number of perseverative errors
Arm/Group | Buspirone Plus Methylphenidate | Placebo for Buspirone Plus Methylphenidate
Number analyzed (Participants) | 20 | 20
number of perseverative errors | 10.88235 (8.305739) | 14.69598 (16.61123)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Buspirone: week 1: Buspirone 30 mg BID weeks 2-3: Buspirone 45 mg BID
  Buspirone: week 1 = 30 mg BID weeks 2-3 = 45 mg BID
- Placebo: week 1: Placebo BID weeks 2-3: Placebo BID
  Placebo: week 1 = placebo BID weeks 2-3 = placebo BID
Arm/Group | Buspirone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=20) | Placebo (N=20)
Elevated Blood pressure (transient) (Cardiac disorders) | 0 (0) | 1 (1)
Upset stomach/nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes